CLINICAL TRIAL: NCT07059533
Title: Non-invasive Brain Stimulation to Enhance the Effects of Training in Healthy Old and Patients With Focal Brain Lesions
Brief Title: Training in Combination With Non-invasive Brain Stimulation
Acronym: TrainStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friedhelm Hummel (Other)
Responsible Party: Sponsor-Investigator, Friedhelm Hummel, Full professor, Ecole Polytechnique Fédérale de Lausanne
Organization: Ecole Polytechnique Fédérale de Lausanne (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2017-00301
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Motor Skill Acquisition in Healthy Older Adults
Keywords: Non-invasive brain stimulation; Transcranial direct current stimulation
MeSH Terms: interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Intervention Model Description: We randomly assigned participants to receive either real or placebo stimulation
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): anodal transcranial direct current stimulation
  Interventions: Other: Verum
- Placebo (Placebo Comparator): 40 seconds of stimulation delivered at the beginning of training (with 8 seconds ramp-up and 5 seconds ramp-down times)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Verum — anodal transcranial direct current stimulation: 20 minutes of stimulation with 1 mA (ramp-up/ramp-down times of 8 seconds)
  Arms: Verum
Other: Placebo — anodal transcranial direct current stimulation with 40 seconds of stimulation delivered at the beginning of training (with 8 seconds ramp-up and 5 seconds ramp-down times)
  Arms: Placebo

SUMMARY:
The goal of this study is to investigate the impact of non-invasive brain stimulation on motor skill acquisition in healthy individuals. Participants performed a motor task with non-invasive brain stimulation applied over the area of the brain where movements were controlled. The study compared motor skill performance between with the active stimulation and the placebo stimulation.

DETAILED DESCRIPTION:
This study implemented a randomized, double-blinded, and sham-controlled design, investigating the effects of non-invasive brain stimulation on motor skill acquisition in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* age equals to or over 18 years old
* absence of major neurological, psychiatric and physical impairment, with normal or corrected to normal vision
* right handed
* in good general health

Exclusion Criteria:

* professional musicians/stenotypist
* unable to consent
* unable to perform the task as required (instructions and setup)
* exclusion criteria for magnetic resonance imaging (MRI), transcranial electrical stimulation (tES), transcranial magnetic stimulation (TMS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Motor performance | From the start of the practice to the end of training at 5 days (and follow up on the 10th day and 60th day)
  Replication of a nine-digit sequence displayed on a screen, as quickly and as accurately as possible, using the left hand

CONTACTS AND LOCATIONS:
Locations (1):
- Campus Biotech, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided